CLINICAL TRIAL: NCT02996981
Title: Do Cranberry Juice Capsules Reduce the Risk of Urinary Tract Infections in Patients With Indwelling Urinary Catheters Following Urogynecologic Surgery?
Brief Title: Cranberry Effect on Urinary Tract Infections
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 16-087
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Results first posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2022-10

CONDITIONS: Urinary Tract Infections
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cranberry group: Patients underwent pelvic floor gynecologic surgery performed by a physician at Cincinnati Urogynecology Associates, TriHealth Inc between April 2016 and September 2016 and discharged home with an indwelling urinary catheter following the surgery. This group of people had cranberry juice capsules prescribed.
- No cranberry group: Patients underwent pelvic floor gynecologic surgery performed by a physician at Cincinnati Urogynecology Associates, TriHealth Inc between April 2015 and September 2015. This group of people did not have cranberry juice capsules prescribed.

SUMMARY:
This is a retrospective chart review using Electronic Privacy Identification Center (EPIC) database to determine if the addition of cranberry juice capsules to our discharge medication regimen for patients discharged home with an indwelling urinary catheter following pelvic floor gynecology surgery reduced the incidence of UTI.

DETAILED DESCRIPTION:
The incidence of urinary tract infection (UTI) in women undergoing pelvic floor gynecologic surgery is high, ranging from 10-64%. A recent randomized trial showed that cranberry juice capsules significantly reduced the incidence of UTI in patients undergoing elective gynecologic surgery (19% vs 38%; odds ratio 0.38 with confidence interval 0.19-0.79).

Cranberry juice capsules were incorporated into the standard practice of Cincinnati Urogynecology Associates, TriHealth Inc in mid-March 2016. Currently, all patients who undergo pelvic floor gynecologic surgery and are discharged from the hospital with an indwelling urinary catheter postoperatively are prescribed cranberry juice capsules to reduce the risk of UTI.

The purpose of this study is to determine if the addition of cranberry juice capsules to the discharge medication regimen for patients discharged home with an indwelling urinary catheter following pelvic floor gynecology surgery significantly reduced the incidence of UTI, compared to a separate cohort that did not have cranberry prescribed.

ELIGIBILITY:
Inclusion Criteria:

* Underwent pelvic floor gynecologic surgery between April 2015 and September 2015, and April 2016 and September 2016
* Required indwelling urinary catheter use upon discharge from the hospital.

Exclusion Criteria:

* Intraoperative bladder injury, fistula repair, urethral diverticulectomy, or any other need for prolonged catheterization
* Complications in the 2 weeks following surgery requiring reoperation and subsequent catheter use
* Allergy to cranberry or its components
* Failure to present for both the two-week and six-week postoperative office visit

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent pelvic floor gynecologic surgery (for the indication of pelvic organ prolapse or stress urinary incontinence) performed by a physician at Cincinnati Urogynecology associates, TriHealth Inc between April 2015 and September 2015, and April 2016 and September 2016
Sampling Method: Non-Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2016-11-21; Primary Completion 2017-07-14 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pauls, MD, Principal Investigator — TriHealth - Cincinnati Urogynecology Associates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shatkin-Margolis A, Warehime J, Pauls RN. Cranberry Supplementation Does Not Reduce Urinary Tract Infections in Patients With Indwelling Catheters After Pelvic Reconstructive Surgery. Female Pelvic Med Reconstr Surg. 2018 Mar/Apr;24(2):130-134. doi: 10.1097/SPV.0000000000000507. PMID 29474286

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cranberry Group | No Cranberry Group
Started | 96 | 71
Completed | 96 | 71
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cranberry Group | No Cranberry Group | Total
Number analyzed (Participants) | 96 | 71 | 167
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.28 (14.10) | 59.62 (15.29) | 60.00 (14.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 71 | 167
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 86 | 64 | 150
  African American | 6 | 4 | 10
  Asian | 1 | 1 | 2
  Hispanic | 3 | 0 | 3
  Other | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 96 | 71 | 167

OUTCOME MEASURES:

1. Primary Outcome: The Incidence of UTI
Time Frame: within 6 weeks postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Cranberry Group | No Cranberry Group
Number analyzed (Participants) | 96 | 71
Participants | 66 | 54
Statistical Analysis 1: Comparison: Cranberry Group vs No Cranberry Group; Test type: Superiority; p = 0.299, Chi-squared; df=1

ADVERSE EVENTS:
Time Frame: From time of surgery to 12 weeks after surgery
Arm/Group | Cranberry Group | No Cranberry Group
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/71
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/71
Other Adverse Events (participants affected / at risk) | 0/96 | 0/71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-04): https://cdn.clinicaltrials.gov/large-docs/81/NCT02996981/Prot_SAP_000.pdf